CLINICAL TRIAL: NCT07346079
Title: A Randomized, Multicenter, Double-blind, Efficacy and Safety Study of 2 Dose Levels of Purified Cortrophin® Gel in Patients With Acute Gouty Arthritis Flares
Brief Title: Purified Cortrophin® Gel Efficacy and Safety Study of 2 Dose Levels in Patients With Acute Gout Flares
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ANI Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Hyon Choi, Physician Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025P001469
Record Dates: First submitted 2025-12-19; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Gout Arthritis; Gout Flare; Gout
MeSH Terms: conditions — Arthritis, Gouty; Gout

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Purified Cortophin Gel 40 U (Experimental): Patients in this arm will receive the 40 U dose at Day 0
  Interventions: Drug: Purified Cortophin Gel, 40 U
- Purified Cortophin Gel 80 U (Experimental): Patients in this arm will receive the 80 U dose at Day 0
  Interventions: Drug: Purified Cortophin Gel 80 U

INTERVENTIONS:
Drug: Purified Cortophin Gel, 40 U — This will be the 40 U dose of the purified Cortophin Gel
  Arms: Purified Cortophin Gel 40 U
Drug: Purified Cortophin Gel 80 U — This will be the 80 U dose of the purified Cortophin Gel
  Arms: Purified Cortophin Gel 80 U

SUMMARY:
This is a randomized, multicenter, double-blind, single administration study to investigate the efficacy and safety of 2 dosing regimens of Purified Cortrophin® Gel in the treatment of an acute gouty arthritis flare.

The study consists of three periods: an optional pre-screening period, a double-blind treatment period, and a 7-day follow-up period.

The treatment period is double-blind, and the patients will be randomized to treatment with 40 U Purified Cortrophin® Gel or 80 U Purified Cortrophin® Gel in a 1:1 ratio. Purified Cortrophin® Gel will be administered once (either subcutaneously or intramuscularly) on the first visit (Day 0; Visit 1) and surveyed after 24 hours (Day 1), 48 hours (Day 2), and 72 hours (Day 3; Visit 2) as well as on Day 7.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in this study
* Male and female patients, aged 18-85 years
* Meeting the 2015 Gout classification criteria of the ACR/EULAR collaborative initiative
* Onset of current acute gout flare within 5 days prior to study entry
* Body mass index of less than or equal to 45 kg/m2
* Baseline pain intensity ≥ 50 mm on the 0-100 mm visual analog scale (VAS)
* History of ≥ 1 gout flares within the 12 months prior to study entry
* The patient meets at least one of the following criteria for both NSAIDs and colchicine treatment options:
* Minimum of one episode of being intolerant, or unresponsive to the treatment, see Appendices 2-4.
* The investigator deems the patient is either contraindicated or inappropriate for the treatment. Inappropriateness could be due to anticipated changes in patient status (i.e., such as worsening of comorbidities or use of concomitant medication), see Appendices 2-4.
* Patients must be willing and capable of using an electronic device (e.g., cellphone) and must have access to a cellphone to be able to complete surveys.

Exclusion Criteria:

* Patients with scleroderma, osteoporosis, active or recurrent bacterial, fungal or viral infections, ocular herpes simplex, recent surgery (within 2 weeks prior to randomization or have an unhealed operation wound(s)), history of or the presence of a peptic ulcer, uncontrolled congestive heart failure, uncontrolled hypertension, uncontrolled diabetes type 1 or 2, or sensitivity to proteins derived from porcine sources.
* Patients with primary adrenocortical insufficiency or adrenocortical hyperfunction.
* Rheumatoid arthritis, evidence or suspicion of infectious/septic arthritis, or other acute inflammatory arthritis.
* Polyarticular gouty arthritis involving more than 4 joints.
* Participation in another concurrent investigational study within 30 days of randomization or has taken an investigational drug within five times the half-life of that investigational drug has passed.
* Previous inclusion in this study.
* Presence of severe renal function impairment: estimated creatinine clearance <30 mL/min/1.73m2 (CKD stages 4 and 5).
* Uncontrolled clinically significant hematologic, CNS, hepatic, pulmonary, gastrointestinal, metabolic, or endocrine disease as deemed by the investigator.
* Presence of any medical or psychological condition or laboratory result that might create risk to the patients (or interfere with the patient's ability to comply with the protocol requirements, or to complete the study) in the opinion of the investigator.
* Prior or current treatment with any ACTH product.
* Pregnant or nursing (lactating) women. Women of childbearing age are required to be using an acceptable method of contraception.
* Patients taking urate-lowering therapy had to be on a stable dose and regimen for ≥2 weeks before entering the study and remain on a stable dosage and regimen for at least 1 week after Purified Cortrophin® Gel.
* Use of specified pain relief medications or biologics (including glucocorticoids, narcotics, paracetamol/acetaminophen, NSAIDs, colchicine, IL-blockers and tumor necrosis factor [TNF] inhibitors) within specified periods (see Appendix 5) prior to randomization.

  * Vaccination within 30 days prior to study enrollment and during the study period.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in gout pain intensity from baseline in target join to 72 hours post-injection | From baseline to Day 3/Visit 2
  Change in gout pain intensity from baseline in the target joint following PCG administration measured by Visual Analog Scale (VAS) at 72 hours post-injection (Day 3; Visit 2).
  Patients will score their pain intensity in the joint most affected at baseline (i.e., the index joint) on a 0-100 mm visual analogue scale (VAS), ranging from no pain (0) to unbearable pain (100).

SECONDARY OUTCOMES:
Change in gout pain from baseline in target joint at Day 1 | From baseline to Day 1
  Change in gout pain intensity from baseline in the target joint following Purified Cortrophin® Gel administration measured by Visual Analog Scale (VAS) at Day 1 (24 hours post-injection).
  Minimum value: 0 Maximum value: 10
  Higher score indicates worse outcome.
Change in gout pain intensity from baseline in target joint to Day 2 | From baseline to Day 2
  Change in gout pain intensity from baseline in the target joint following Purified Cortrophin® Gel administration as measured by Visual Analog Scale (VAS) at Day 2 (48 hours post-injection).
  Minimum value: 0
  Maximum value: 10
  Higher score indicates worse outcome.
Change in pain intensity timeline at baseline, 24 hours, 48 hours, 72 hours, and Day 7 post-injection. | From baseline to Day 7
  Change in pain intensity timeline at baseline, 24 hours, 48 hours, 72 hours, and Day 7 post-injection.
Time to onset of effect (≥20% change from baseline pain intensity on VAS). | From baseline to end of study (Day 7)
  Time to onset of effect (≥20% change from baseline pain intensity on VAS).
Time to response (≥50% change from baseline pain intensity on VAS). | From baseline to end of study (Day 7)
  Time to response (≥50% change from baseline pain intensity on VAS).
Patient Global Self-Assessment to treatment: (24 hours, 48 hours, 72 hours, and Day 7 post-injection). | From baseline to end of study (Day 7)
  Patient Global Self-Assessment to treatment: (24 hours, 48 hours, 72 hours, and Day 7 post-injection).
  4 - Excellent 3 - Good 2 - Acceptable
  1 - Slight 0 - Poor
  Lower scores indicate worse outcomes.
Physician assessment of inflammatory signs: (baseline [Day 0; Visit 1], 72 hours [Day 3; Visit 2]) | From baseline to end of study (Day 7)
  Physician assessment of inflammatory signs: (baseline [Day 0; Visit 1], 72 hours [Day 3; Visit 2])
  * Physician assessment of joint tenderness
    0 - No pain
    1. - Mild/patient there is pain when touched
    2. - Moderate/patient states there is pain and winces
    3. - Severe/patient states there is pain, winces and withdraws.
  * Physician assessment of joint swelling
    0 - No swelling
    1. - Mild swelling/palpable
    2. - Moderate swelling/visible
    3. - Severe swelling/bulging beyond the joint margins
  * Physician assessment of erythema
  Absent or Present
  o Physician assessment of target joint range of motion
  0 - Normal
  1. - Mildly restricted
  2. - Moderately restricted
  3. - Severely restricted
  4. - Immobilized
  The above answers will be totaled - minimum value: 0, max: 12. Higher values indicate worse outcomes.
Physician assessment of local tolerability at injection site (at 72 hours post-injection). | Day 3 (Visit 2)
  Physician assessment of local tolerability at injection site (at 72 hours post-injection)
  Notes presence of redness, swelling, pain, bruising, itching (no numerical values).
Use of rescue medication (up to 72-hours post-injection). | From baseline to Day 3/Visit 2
  Use of rescue medication (up to 72-hours post-injection).
Safety assessment - AEs, SAEs | From baseline to end of study (Day 7)
  Notes presence, description, duration of an AE, and whether the AE is serious.
Safety Assessment - Vital Signs | Day 1 Visit and Day 3 Visit
  Height and Weight will be collected, and used to calculate the participant's BMI
Safety Assessment - Laboratory Measurements | Day 1 and Day 3
  Biochemistry:
  Aspartate aminotransferase (AST) Alanine aminotransferase (ALT) Total bilirubin (if >upper limit of normal also conjugated and non-conjugated bilirubin) Alkaline phosphatase (ALP） Prothrombin Time/International Normalized Ratio (PT/INR)‡¥§ Albumin Cholesterol (total, LDL, and HDL) Triglycerides Creatinine◊§ Sodium (Na) Potassium (K) Ferritin Erythrocyte sedimentation rate Uric acid Glucose*¥ HbA1c Troponin T C-reactive protein (CRP) Serum amyloid A (SAA) Calcium Magnesium
  Hematology:
  Hemoglobin Hematocrit White blood cells Differential blood count Thrombocytes
  Urine analysis:
  Albumin U-erythrocytes
  Abnormal test findings, if changed significantly from baseline will be noted. Minimum and maximum values, as well as indications of higher or lower values vary depending on the test.

OTHER OUTCOMES:
Levels of inflammatory markers (baseline [Day 0; Visit 1], 72 hours [Day 3; Visit 2]) | From baseline to Day 3/Visit 2
  Levels of inflammatory markers (baseline [Day 0; Visit 1], 72 hours [Day 3; Visit 2])
  * C-reactive protein
  * Serum amyloid A
Change from baseline in health-related quality-of-life Gout Attack Intensity Score (GAIS) at Day 0 (Visit 1) and at Day 3 (72-hours post-injection; Visit 2) (19). | From baseline to Day 3/Visit 2
  Change from baseline in health-related quality-of-life Gout Attack Intensity Score (GAIS) at Day 0 (Visit 1) and at Day 3 (72-hours post-injection; Visit 2) (19).
  1. How much pain is your gout causing you today? (color in one box completely)
     * 1 No pain
     * 2 Mild pain
     * 3 Moderate pain
     * 4 A lot of pain
     * 5 Extreme pain
  2. How tender to the touch are the gout-affected parts of your body today? (colour in one box completely)
     * 1 Not tender
     * 2 Slightly tender
     * 3 Fairly tender
     * 4 Very tender
     * 5 Extremely tender
  3. How swollen are the gout-affected parts of your body today? (colour in one box completely)
     * 1 Not swollen
     * 2 Somewhat swollen
     * 3 Fairly swollen
     * 4 Very swollen
     * 5 Extremely swollen
  The answers across all three questions will be totaled, with higher scores indicating worse outcomes. Minimum value: 3, maximum value: 15

CONTACTS AND LOCATIONS:
Overall Officials: Hyon K Choi, MD, DrPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared with the sponsor.